CLINICAL TRIAL: NCT04447001
Title: Improving Balance for Older Adults: Disseminating Tai Chi Fundamentals Through Community Organizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0897; A561000 (Other: University of Wisconsin, Madison); PHARM/PHARMACY/PHARMACY (Other: University of Wisconsin, Madison)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Older Aged Adults; Balance
Keywords: Tai Chi

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to immediately begin short 6-week modified tai chi course along with a personal home practice plan to receive greater Tai chi dose(session 1) or complete a 8-week wait (wait-list control). Wait-list group will be receiving Tai-chi prime intervention after 8 weeks wait time (session-2).
  In addition to the pre-post tests of TCF sessions to explore TCF effectiveness, pre-test scores for session 2 are compared to post-test scores of session 1 participants since both are collected at nearly the same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi Prime (TCP)-session 1 (Experimental): This arm will receive Tai chi prime as an intervention. TCP is a combination of two components: (a) Tai-chi fundamental Adapted Program, and (b) home practice coaching.
  Interventions: Behavioral: Tai-chi prime (TCP)
- Wait list control-session 2 (No Intervention): Wait-list group will be receiving Tai-chi prime intervention after 8 weeks wait time. At week 7, pre-test measures from wait-list group will be used as a control and compared with the post intervention measures of the experimental group.

INTERVENTIONS:
Behavioral: Tai-chi prime (TCP) — TCP is a 6-week twice-weekly simplified tai chi class of 1.5 hr per session with two components: (a) Tai-chi fundamental Adapted Program, and (b) home practice coaching.
  Arms: Tai Chi Prime (TCP)-session 1

SUMMARY:
This study will evaluate how best to disseminate and implement Tai Chi Fundamentals® (TCF) in community settings for older adults with balance problems. TCF is a program designed for older adults with pain and physical limitations to enhance balance, coordination, strength and endurance. Investigator will evaluate program implementation including Aging and Disability Resource Center (ADRC) uptake, reach, feasibility, teaching fidelity, and exercise adherence and also collect outcomes including leg strength, balance, walking ability and executive function before and after the 6-week session. The final product of this study will be recommendations to address key barriers and facilitators for implementation of TCF by community organizations serving older adults.

The primary aim for this study is to evaluate the program implementation. This is not an efficacy study. Within the limits of a Dissemination and Implementation grant budget, Investigators do take advantage of a natural experiment even if it is not the primary aim of this study. By doing so investigators plan to establish the feasibility of this multi-site data collection plan for future studies. Based on the study settings, study team will get a chance to explore the effect of TCF in real world settings since two sessions can be held in a fall season and a spring season. In addition to the pre-post tests of TCF sessions to explore TCF effectiveness, pre-test scores for session 2 are compared to post-test scores of session 1 participants since both are collected at nearly the same time. The larger sample will be for the within group pre-post comparison analyses. This will be a valuable opportunity to test data collection procedures for future trials.

ELIGIBILITY:
Inclusion Criteria:

* being 65 years and older
* dwelling independently in the community
* agreeing to be randomized
* reporting a fall (to the ground or lower level in the last year or having a strong fear of falling.

Exclusion Criteria:

* using a walker indoors
* having a terminal illness
* being hospitalized or in a nursing home in the past 2 months
* anticipated absence from two tai chi sessions and
* receiving physical therapy or a community course or balance exercise program for falls prevention in the prior 2 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of participants retention | 7 week (for session 1) ,7 week ( for session 2)
  Rate of participant retention in 2 sessions of TCP
Number of days participants practiced Tai-chi at home | 7 week (for session 1) , 7 week( for session 2)
  Participants will report the average time they are practicing Tai-chi every day at home

SECONDARY OUTCOMES:
Change in the time taken to complete 'Trail Making Test Part B' | baseline for session 1, 7 weeks (post test for session 1) and 7 weeks (pretest for session 2)
  The Trail Making Test(TMT) is a neuropsychological test of visual attention and task switching. In TMT, the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The time taken to complete the test being used as the primary performance metric.
Change in Activities-specific Balance Confidence (ABC) Scale score | baseline for session 1, 7 weeks (post test for session 1) and 7 weeks (pretest for session 2)
  The ABC scale is a self- report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness.
  ABC is an 11-point scale and ratings should consist of whole numbers (0-100) for each item. Participants will indicate their level of confidence in doing an activity without losing balance or becoming unsteady by choosing one of the percentage points on the scale from 0%-100%. Total the ratings (possible range = 0 to 1600) and divide by 16 to get each participant's ABC score.
  Scores lower than 50 indicate a low level of functioning, scores above 50 but below 80 indicate a medium level, and those over 80 indicate a high level of functioning.
Change in the static balance as measured by Single-leg Balance | baseline for session 1, 7 weeks (post test for session 1) and 7 weeks (pretest for session 2)
  Static balance is the ability to maintain the body in some fixed posture.
Change in time taken to complete TUG (Timed Up and Go) test | baseline for session 1, 7 weeks (post test for session 1) and 7 weeks (pretest for session 2)
  TUG test is a test of mobility and gait. Participant will timed for the following TUG test
  * Participants will be asked to sit back in a standard chair and identify a line 3 meters, or 10 feet away.
  * At 'Go' participant will stand up from the chair.
  * Walk to the line on the floor at your normal pace.
  * Turn.
  * Walk back to the chair at your normal pace.
  * Sit down again.
  Time taken from start to finish will be measured in seconds.
  An older adult who takes ≥12 seconds to complete the TUG is at risk for falling.
Change in the time taken to hold tandem stands in the 4-stage balance test | baseline for session 1, 7 weeks (post test for session 1) and 7 weeks (pretest for session 2)
  4 stage balance test consists of four standing positions that get progressively harder to maintain.
  instructor will describe and demonstrate each position to the participant.Then the instructor will stand next to the participant, hold their arm,and help them assume the correct position. When the participant will be steady, let go, and time how long they can maintain the position. Instructor will be ready to assist the participant if they lose their balance.
  If the participant can hold a position for 10 seconds without moving their feet or needing support, instructor can ask to go on to the next position. If not, test will be stopped.
  Participants should not use an assistive device (cane or walker) and they should keep their eyes open.
  Participants (older adults) who cannot hold the tandem stand for at least 10 seconds will be at increased risk of falling.
Change in the 'number of times the participant comes to a full standing position in 30 seconds' | baseline for session 1, 7 weeks (post test for session 1) and 7 weeks (pretest for session 2)
  The 30 Second Chair Stand Test can help to indicate if a patient is at risk of falling. Purpose of this test is to test the strength and endurance.
  Instructions to the participant:
  * Sit in the middle of the chair.
  * Place each hand on the opposite shoulder crossed at the wrists.
  * Place your feet flat on the floor.
  * Keep your back straight and keep your arms against your chest.
  * On "Go", rise to a full standing position and then sit back down again.
  * Repeat this for 30 seconds.
  On "Go" timer starts.
  Number of times the participant comes to a full standing position in 30 seconds will be recorded.
  If the participant is over halfway to a standing position when 30 seconds have elapsed, it will be counted as stand.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Chewning, PhD, Principal Investigator — University of Madison
Locations (3):
- United States (3):
  - Aging and Disability Resource Center (ADRC), La Crosse, Wisconsin
  - Goodman Community Center, Madison, Wisconsin
  - Milwaukee County Department on Aging, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chewning B, Hallisy KM, Mahoney JE, Wilson D, Sangasubana N, Gangnon R. Disseminating Tai Chi in the Community: Promoting Home Practice and Improving Balance. Gerontologist. 2020 May 15;60(4):765-775. doi: 10.1093/geront/gnz006. PMID 30811543